Official Title: Multicenter, Open-label Active-controlled Randomized Study of Efficacy and

Safety of Ferrum Lek® (Iron (III) Hydroxide Polymaltosate), 100 mg Chewable Tablets (Lek d.d., Slovenia) Compared With Maltofer® (Iron (III) Hydroxide Polymaltosate), 100 mg Chewable Tablets (Vifor S.A., Switzerland), in Treatment of Patients With Mild and Moderate Iron-deficiency Anaemia

NCT Number: NCT03993288

**Document Date:** Statistical Analysis Plan Version 1.0: 06 April 2020

| /Logotype: Research/ | STATISTICAL ANALYSIS PLAN |
|----------------------|---------------------------|

## **Statistical Analysis Plan**

| Sponsor | Sandoz CJSC |
|---|---|
| | A multicenter, open-label, randomized, active-controlled |
| | study to evaluate the efficacy and safety of Ferrum Lek® |
| | (iron (III) hydroxide polymaltosate), 100 mg chewable tablets |
| Protocol title | (Lek d.d., Slovenia), as compared to Maltofer® (iron (III) |
| | hydroxide polymaltosate), 100 mg chewable tablets |
| | (Vifor S.A., Switzerland), in subjects with mild and moderate |
| | iron deficiency anemia |
| Protocol No. | TE 005 FER CHT |

| Author | |
|-----------------------------------|---------------|
| Statistical Analysis Plan version | 1.0 |
| Date of version | April 6, 2020 |

## STATISTICAL ANALYSIS PLAN

## Approved by

| Full name | Position | Signature | Date |
|-----------|----------|-------------|---------------|
| | | /Signature/ | April 6, 2020 |
| | | /Signature/ | April 6, 2020 |
| | | /Signature/ | April 6, 2020 |
| | | /Signature/ | April 6, 2020 |

## **Document history**

| Version | Reason for change | Date |
|---------|-------------------|---------------|
| 1.0 | Original document | April 6, 2020 |

## STATISTICAL ANALYSIS PLAN

## **Table of contents**

| 1. | | on | |
|------------|----------------|------------------------------------------|----|
| 2. | Study obj | ectives and design | 7 |
| | 2.1. Stud | y objectives | 7 |
| | | Primary objective | |
| | 2.1.2. | | |
| | 2.2. Stud | y design | |
| | | tudy design flowchart | |
| | | n of visits | |
| | | ple size | |
| 3. | | nalysis values | |
| - | | eral assumptions and baseline conditions | |
| | | essing missing data | |
| 4 | | ticipants | |
| ٠. | | ent distribution | |
| | | y population | |
| | 4.3.1. | Safety population | |
| | | ITT population receiving treatment | |
| | 4.3.3. | Per protocol set | |
| 5. | | phics and baseline characteristics | |
| <i>5</i> . | | ant therapy | |
| 0. | | nitted concomitant therapy | |
| | 6.1. Felli | ibited concomitant therapy | 15 |
| 0 | | nalysis | |
| ٥. | | nary endpoint analysis | |
| 0 | | lysis of the secondary endpoint | |
| 9. | • | alysis | |
| | | erse events | |
| 1.0 | | er safety endpoints | |
| | | ry analysis | |
| | | nalysis | |
| Ap | | able layouts | |
| | | RY ENDPOINTS | |
| | | ORY RESULTS | |
| | | inalysis | |
| | | inalysis statistical test | |
| | | inalysis, categorical variables | |
| | | matology 1 | |
| | | matology 2 | |
| | | ematology 3 | |
| | | ematology 4 | |
| | | ematology, statistical test 1 | |
| | | ematology, statistical test 2 | |
| | | Iematology, statistical test 3 | |
| | | lematology, statistical test 4 | |
| | | hysiological data | |
| | | hysiological data, statistical test | |
| | | hysiological data, categorical data | |
| | | iochemistry 1 | |
| | | iochemistry 2 | |
| | | iochemistry 3 | |
| | | iochemistry, statistical test 1 | |
| | | iochemistry, statistical test 2 | |
| | | iochemistry, statistical test 3 | |
| | <b>ADVERSE</b> | E EVENTS | 65 |

#### STATISTICAL ANALYSIS PLAN /Logotype: Research/

| Table 1. Adverse events reported in the study | 65 |
|---|---|
| Tables N. Is the adverse event ongoing?/ Relatedness to the medicinal product/ Dose a | djustment or temporary |
| withdrawal of the IMP/ Complete withdrawal of the IMP/ Prescribing a concomitant | medicinal product/ |
| Prescribing non-drug therapy/ Patient admission to hospital or hospitalization prolon | gation/ Based on an AE/ Is it |
| an SAE?/ Leads to death/ Threatens life/ Requires admission to hospital or hospitaliza | ation prolongation/ Leads to |
| permanent or significant incapacity for work or disability | 66 |

## STATISTICAL ANALYSIS PLAN

## List of abbreviations and definitions of terms

| ANOVA | Analysis of variance |
|---|---|
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HFE | Hemochromatosis gene |
| ICH | The International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use |
| ITT | Intention-to-treat |
| LD100 | Lethal dose, the average dose of the substance in milligrams per kilogram of live weight, which causes the death of 100% of experimental animals |
| LD50 | Half-lethal dose, the average dose of the substance in milligrams per kilogram of live weight, which causes the death of 50% of experimental animals |
| MLE | Maximum likelihood estimation |
| PP | Per protocol |
| BP | Blood pressure |
| ALT | Alanine aminotransferase |
| JSC | Joint-stock company |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical (classification system) |
| VAS | Visual analog scale |
| HIV | Human immunodeficiency virus |
| IUS | Intrauterine system |
| IUD | Intrauterine device |
| Hb | Hemoglobin |
| GOST | State standard |
| GOSTR | State Standard of Russia |
| DBP | Diastolic blood pressure |
| ID | Iron deficiency |
| CI | Confidence interval |
| DMPO | 5,5-Dimethyl-1-pyrroline-N-oxide |
| IDA | Iron-deficiency anemia |
| GI | Gastrointestinal |
| GI tract | Gastrointestinal tract |

| CRF | Case record form |
|---|---|
| CRO | Contract research organization |
| LDL | Low-density lipoprotein |
| МоН | Ministry of health |
| MIC | Minimum inhibitory concentration |
| ICD | International Classification of Diseases |
| GCP | Good Clinical Practice |
| IEC | Independent ethics committee |
| AE | Adverse event |
| SmPC | Summary of Product Characteristics |
| PVC | Polyvinyl chloride |
| IHPC | Iron (III) hydroxide polymaltose complex |
| IPC | Iron polymaltose complex |
| PND | Postnatal days |
| PCR | Polymerase chain reaction |
| RMSAH/ | The Russian Medical Society on Arterial Hypertension/ The Russian Society of |
| RSC | Cardiology |
| ITP | Iron transport proteins 1 and 2 |
| RE | Reticuloendothelial (cells) |
| RES | Reticuloendothelial system |
| SBP | Systolic blood pressure |
| SAE | Serious adverse event |
| SOD | Superoxide dismutase |
| SOP | Standard operating procedure |
| TF | Transferrin |
| TfR | Transferrin receptor |
| FL | Federal law |
| Full name | First name, Patronymic, Last name |
| CNS | Central nervous system |
| Ср | Ceruloplasmin |
| RR | Respiration rate |
| HR | Heart rate |
| ECG | Electrocardiography |

### STATISTICAL ANALYSIS PLAN

#### 1. Introduction

This study is planned and carried out to demonstrate the non-inferiority and safety of Ferrum Lek® (iron (III) hydroxide polymaltosate), 100 mg chewable tablets (Lek d.d., Slovenia), compared to MALTOFER® (Vifor S.A., Switzerland), in subjects with mild and moderate iron deficiency anemia.

The objective of this Statistical Analysis Plan is more detailed, compared to Section 9 of the study protocol, description of the main principles of the protocol-based statistical analysis, description of the primary and secondary endpoints analysis methods as well as other data obtained during the study.

This Plan stipulates for conformance of the scheduled and conducted statistical analysis to the study protocol, including the definition of the analysis data sets, transformations and calculations for the endpoints, observations quantity needed, etc.

### 2. Study objectives and design

#### 2.1. Study objectives

#### 2.1.1. Primary objective

To demonstrate non-inferior therapeutic efficacy of Ferrum Lek® by evaluating its effect on blood hemoglobin levels (g/L) when taken as 2 tablets (200 mg) per day for 12 weeks in subjects with mild to moderate iron deficiency anemia versus 2 tablets (200 mg) per day of MALTOFER® administered over the same period.

#### 2.1.2. Secondary objectives

To evaluate the safety of Ferrum Lek® with 2 tablets (200 mg) per day versus MALTOFER® with 2 tablets (200 mg) per day by evaluating the rates, characteristics, severity of AEs, and their relation to the prescribed treatment.

#### 2.2. Study design

This study is a multicenter, randomized, open-label, prospective, comparative, phase III, parallel-group, active control study conducted in the Russian Federation.

The eligible and ineligible subjects will be randomized into two treatment groups at the ratio of 1:1.

The subjects in the first group (168 subjects) will receive 2 tablets daily (200 mg) of Ferrum Lek® chewable tablets, during or right after meals; the daily dose should be administered once daily (as a single dose). The subjects in the second group (168 subjects) will receive 2 tablets daily (200 mg) of MALTOFER® chewable tablets, during or right after meals; the daily dose should be administered once daily. Subjects will take the medicinal products daily for 12 weeks and fill out a diary (see Appendix 17.1), where they will register administration of the study medicinal products and concomitant therapy.

### STATISTICAL ANALYSIS PLAN

All subjects will undergo a complete blood count and blood biochemistry. Therapy under investigation also includes an interim Visit 2 (Day  $29 \pm 2$ ), Visit 3 (Day  $57 \pm 2$ ), and final Visit 4 ( $84 \pm 2$ ). After the final visit, a subject's participation in the study shall be terminated, and further treatment shall be performed by a consulting physician.

The study design is depicted in Figure 1.

#### 4.2.6. Study design flowchart



Figure 1. Study design flowchart

#### **Study duration**

The total duration of the study will be no more than 12 months, including enrollment (9 months), treatment (3 months), and follow-up (by phone) 14 days after the completion of the active treatment period.

Description of visits

#### 4.2.9.1. Visit 0 (screening, days -7...-1)

#### Visit objectives:

- Signing of the informed consent;
- Assessment of the inclusion/exclusion criteria;

- Collection of demographic and anthropometric data;
- Collection of medical history data on iron deficiency anemia and significant concomitant diseases;
- Physical examination, blood pressure and heart rate measurement;
- Laboratory tests:
  - o Urinalysis [general properties (color, pH, specific gravity, protein) and sediment microscopy];
  - Urine pregnancy test;
  - o HIV antibody test, except for subjects who had an HIV test within the last 6 months;
  - o Blood biochemistry (total protein, total and conjugated bilirubin, AST, ALT, alkaline phosphatase, creatinine, glucose, CRP);
  - o Complete blood count (hemoglobin level, hematocrit, RBC, PLT, WBC, leucogram, ESR);
  - o Metabolic parameters of iron (serum ferritin and iron level, transferrin, iron transferrin saturation percentage);
  - o Determining blood vitamin B9 (folic acid) and vitamin B12 (cyanocobalamin) levels;
  - o Determining blood TSH and T4 levels;
  - o Creatinine clearance calculation according to the Cockroft-Gault formula;
- Evaluation of the concomitant therapy; Adverse events registration.

#### 4.2.9.2. Visit 1 (randomization/ start of the treatment, Day 1)

#### **Visit objectives:**

- Assessment of the inclusion/exclusion criteria;
- Randomization;
- Start of the treatment with the investigational medicinal product;
- Hand-out of the patient diary (Appendix 17.1) and instructions on its completion;
- Accounting and dispensing of the investigational medicinal product;
- Evaluation of the concomitant therapy; Adverse events registration.

### 4.2.9.3. Visit 2 (continuation of the treatment, Day $29 \pm 2$ )

#### Visit objectives:

• Physical examination, blood pressure and heart rate measurement;

### STATISTICAL ANALYSIS PLAN

- Metabolic parameters of iron (serum ferritin and iron level, transferrin, iron transferrin saturation percentage);
- Complete blood count (hemoglobin level, hematocrit, RBC);
- Hand-out of the patient diary (Appendix 17.1) and instructions on its completion;
- Check of a patient diary completion and collection of diaries;
- Accounting and dispensing of the investigational medicinal product;
- Evaluation of compliance;
- Evaluation of the concomitant therapy;
- Adverse events registration.

#### 4.2.9.4. Visit 3 (continuation of the treatment, Day $57 \pm 2$ )

#### Visit objectives:

- Physical examination, blood pressure and heart rate measurement;
- Metabolic parameters of iron (serum ferritin and iron level, transferrin, iron transferrin saturation percentage);
- Complete blood count (hemoglobin level, hematocrit, RBC);
- Hand-out of the patient diary (Appendix 17.1) and instructions on its completion;
- Check of a patient diary completion and collection of diaries;
- Accounting and dispensing of the investigational medicinal product;
- Evaluation of compliance;
- Evaluation of the concomitant therapy;
- Adverse events registration.

#### 4.2.9.5. Visit 4 (efficacy and safety assessment, Day $84 \pm 2$ )

#### Visit objectives:

- Physical examination, blood pressure and heart rate measurement;
- Laboratory tests:
  - Urinalysis [general properties (color, pH, specific gravity, protein) and sediment microscopy];
  - Urine pregnancy test;

### STATISTICAL ANALYSIS PLAN

- Blood biochemistry (total protein, total and conjugated bilirubin, AST, ALT, alkaline phosphatase, creatinine, glucose, CRP);
- o Complete blood count (hemoglobin level, hematocrit, RBC);
- Metabolic parameters of iron (serum ferritin and iron level, transferrin, iron transferrin saturation percentage).
- Check of a patient diary completion and collection of diaries;
- Accounting and dispensing of the investigational medicinal product;
- Evaluation of compliance;
- Evaluation of the concomitant therapy;
- Adverse events registration.

#### **4.2.9.6.** Follow-up visit (Visit 5, Day $98 \pm 2$ )

A follow-up visit shall be conducted by phone to find out about the patient's state and any AEs. It will be conducted 14 days after the completion of treatment.

Follow-up visit procedures (by phone):

o Evaluation of adverse events.

In case of adverse events, the patient might be invited to visit the study site.

#### 2.3. Sample size

The sample size was calculated on the basis of the published articles, where the efficacy of iron (III) hydroxide polymaltosate was studied:

- 1) Maltofer, Product Information http://www.aspenpharma.com.au/product\_info/pi/PI\_Maltofer.pdf
- 2) Santiago P. Ferrous versus ferric oral iron formulations for the treatment of iron deficiency: a clinical overview. Scientific World Journal. 2012;2012:846824.
- 3) Geisser P. Safety and efficacy of iron(III)-hydroxide polymaltose complex / a review of over 25 years' experience. Arzneimittelforschung. 2007;57(6A):439-52;
- 4) Toblli JE, Brignoli R. Iron(III)-hydroxide polymaltose complex in iron deficiency anemia/ review and meta-analysis. Arzneimittelforschung. 2007;57(6A):431-8);
- 5) Reinisch W, Staun M, Tandon RK, Altorjay I, Thillainayagam AV, Gratzer C, Nijhawan S, Thomsen LL. A randomized, open-label, non-inferiority study of intravenous iron isomaltoside 1,000 (Monofer) compared with oral iron for treatment of anemia in IBD (PROCEED). Am J Gastroenterol. 2013 Dec;108(12):1877-88.

### STATISTICAL ANALYSIS PLAN

6) Zaim M, Piselli L, Fioravanti P, Kanony-Truc C. Efficacy and tolerability of a prolonged release ferrous sulphate formulation in iron deficiency anaemia: a non-inferiority controlled trial. Eur J Nutr. 2012 Mar;51(2):221-9.

Based on these publications, the hemoglobin levels increased by an average of 8–15 g/L, with SD of up to 15 g/L, following 12 weeks of oral administration of iron (III) hydroxide polymaltosate complex preparations. Since approximately the same efficiency is assumed in both groups, a zero difference in the main efficiency parameter will be used to calculate the sample size. In order to take into account the maximum variability of the primary endpoint variable for the study with sufficient statistical power, the maximum standard deviation value of 15 g/L was used.

The value of 5 g/L was chosen as the non-inferiority cut-off (in accordance with the limit established and justified in the above publications).

Thus, the following assumptions were proposed for calculations:

- 1) It is assumed that changes in the hemoglobin level in the blood (g/L) after 12 weeks of iron deficiency anemia therapy (at the final visit) compared to the initial value (at Screening Visit 0) will be approximately the same in the group receiving the investigational medicinal product and in the group receiving the reference product (i.e., the expected difference between the two groups will be zero).
- 2) A pooled standard deviation for the changes in hemoglobin levels was 15 g/L.
- 3) The non-inferiority margin is 5 g/L.
- 4) The significance level (two-sided, according to the recommendations by the Food and Drug Administration) is 95%, which corresponds to a one-sided type I error of 0.05.
- 5) The study power is 80%, which corresponds to a type II error of 0.20.
- 6) Statistical hypotheses are the demonstration of non-inferiority:

- 7) The ratio between the test and control group sizes is 1:1.
- 8) The interim analysis will be conducted when 70% of the total sample size is reached.
- 9) The O'Brian-Fleming alpha-spending function will be applied with 80% power for the efficiency frontier, which will satisfy the following critical values of the t-test: 2.628 for the intermediate analysis (corresponding to p = 0.005) and 1.976 for the final analysis (corresponding to p = 0.0245).

Calculations were performed using the clinfun package of the R software, in which the calculation of a fixed sample size for interim and final analyses was performed using the group sequential design.

According to the data obtained with the clinfun package, 143 subjects in each group (total: 286 subjects) should complete the study to confirm the hypothesis of non-inferiority. For the interim analysis, data for 200 subjects (100 in each group) that are suitable for analysis should be obtained. Taking into account the frequency of premature discontinuation of the study, which is 15%, it is necessary to randomize 336 people (168 people in each group). Taking into consideration the withdrawal rate based on the results of the screening that equals to 30%, about 480 people should undergo screening to achieve the target level of randomization.

### 3. General analysis values

#### 3.1. General assumptions and baseline conditions

#### Clinical and statistical significance

All the statistical tests within this study will be performed at a 95% confidence level (threshold value p to confirm statistical significance is 0.05).

#### 3.2. Processing missing data

A method of filling in the missing data based on maximum likelihood estimation (MLE) for the primary endpoint will be applied if needed.

The analysis of the rest of endpoint types and other parameters will be performed only on the basis of the available information without filling in the missing data in view of the short duration of the clinical study.

#### 4. Study participants

#### 4.1. Patient distribution

Upon signing of the informed consent for participation in the study, the subjects undergo screening for up to 7 days. The eligible and ineligible subjects will be randomized into two treatment groups at the ratio of 1:1.

Automated randomization sheets will be generated; randomization will be carried out through an electronic CRF system with a randomization module.

Each randomized patient will receive a unique number for the medicinal product dispensing during the study. The patient's number contains R letter and numbers from 001 to 336. Patients numbering does not depend on the study site and is consecutive. In addition to the number, the system will indicate the treatment group to which the patient is randomized. Randomization will be stratified according to two factors: 1) Sex (men vs. women); 2) Hemoglobin level (80–94 g/L versus 95–110 g/L). The randomization number cannot be changed during the study.

The medicinal product is given to the patient according to the information about the treatment group received from the CRF system. Study treatment also cannot be changed in the process of the study.

Serious deviations from the Protocol should be reported as soon as possible to the Sponsor by the site staff and/or CRO and Monitor (if they are at the Site).

The Sponsor must be informed of minor protocol deviations within 10 business days but before the start of the next study period or before the start of the bioanalytical/statistical phase.

Sponsor has the right to terminate the study, and the Investigator has the right to stop subjects recruitment at any time. In the case of premature closing of the center/study, all completed as well as unused CRFs (including unused pages of partially completed CRFs) and other documents (excluding documents that must be kept in the center) must be returned to the Sponsor. Study materials can be destroyed only with the consent of the Sponsor.

#### 4.3. Study population

#### 4.3.1. Safety population

All randomized subjects who received at least one dose of the investigational medicinal product and completed at least one safety parameters evaluation visit. As distinct from ITT population, the TS population will be analyzed depending on actually received treatment (not only prescribed) (in case of difference between the prescribed and received therapies).

#### 4.3.2. ITT population receiving treatment

All randomized subjects who received at least one dose of the investigational medicinal product and completed at least one efficacy parameters evaluation visit.

#### 4.3.3. Per protocol set

All randomized subjects who completed participation in the study in accordance with the protocol (have completed the prescribed period of treatment and follow-up without significant deviations from the protocol).

#### 5. Demographics and baseline characteristics

All the data obtained in the groups before the study therapy initiation (demographic, laboratory, instrumental, and physical examinations data, vital signs, etc.) will be compared between the groups to determine the groups' comparability for analysis.

The Fisher's exact test and  $\chi^2$  (chi-square) will be used to compare the qualitative and serial data, while the t-test or the Mann–Whitney test will be used for the quantitative data (depending on the quantitative data distribution).

To assess the normality of the distribution, the Shapiro-Wilk test will be applied. In the event that any of the initial data reveal the incomparability of the study groups (statistically significant differences in demographic and other initial data between the groups), the analysis of the efficacy and safety parameters will be additionally performed, together with the primary planned analysis, using multi-factor statistics (ANOVA, ANCOVA, or logistic regression analysis depending on the type of the studied parameter), as adjusted for the initial indicator(s) that vary between the groups.

#### 6. Concomitant therapy

#### 6.1. Permitted concomitant therapy

Patients will take medications, which they took before the enrollment, for the treatment of concomitant diseases during the study. Women that take oral contraceptives may continue taking them during the study.

It is permitted and recommended to take vitamins (not containing iron), folic acid, and ascorbic acid by medical prescription as well as adhere to a diet with products rich in iron.

It is not recommended to take non-steroidal anti-inflammatory medicinal products groundlessly, including selective inhibitors of cyclooxygenase, but these medicinal products may be prescribed by the Investigator due to medical indications.

#### **6.2.** Prohibited concomitant therapy

During the study, the enrolled patients must not take the following products:

• prescribed for iron deficiency anemia:

| Pharmacotherapeutic groups | Active substance (INN) |
|-------------------------------------|------------------------|
| Vitamin and mineral supplements | |
| Macro- and microelement supplements | |
| Vitamins and pseudovitamins | Ascorbic acid |

## STATISTICAL ANALYSIS PLAN

| | Dymidavina |
|---|---|
| | Pyridoxine |
| | Riboflavin |
| Vitamin and pseudovitamins in combinations | Multivitamins + Minerals |
| Macro- and microelements | Iron protein succinylate |
| | Hematogen |
| Macro- and microelements in combinations | Ferrous sulfate + Serine + Folic acid |
| Wacro- and inicroelements in combinations | Multivitamins + Minerals |
| | Iron (III) hydroxide polymaltosate complex |
| | Iron (III) hydroxide sucrose complex |
| | Ferrous gluconate |
| | Ferric carboxymaltosate |
| Hematopoiesis-stimulating agents | Iron protein succinylate |
| | Ferrous sulfate |
| | Ferrous fumarate |
| | Ferrous chloride |
| | Cyanocobalamin |
| | Iron (III) hydroxide polymaltosate complex + Folic |
| III | acid |
| Hematopoiesis-stimulating agents in combinations | Ferrous sulfate + Folic acid + Cyanocobalamin |
| Comoniations | Ferrous sulfate + Folic acid |
| | Ferrous fumarate + Folic acid |

and any other substances affecting hematopoiesis (for example, cytostatic agents, interferons, chloramphenicol, streptomycin).

- Other substances that influence hematopoiesis (epoetins, anabolic steroids, etc.)
- Medicinal products that slow iron absorption (antacids, calcium supplements), 2 hours before administration of the investigational products. It is not recommended to drink strong tea and coffee 2 hours before the administration of medicinal products.

During the study, the patients must not undergo physiotherapy or other procedures that potentially affect erythropoiesis (for example, Buteyko breathing).

#### 8. Efficacy analysis

### 8.1. Primary endpoint analysis

• Changes in hemoglobin level (g/L) after 12 weeks of iron deficiency therapy (at the final visit) as compared to baseline (determined at the screening visit) in the study groups.

### STATISTICAL ANALYSIS PLAN

The covariance analysis (ANCOVA) will be used as the main method for assessing the primary endpoint, with the baseline blood hemoglobin level as a covariate, and four fixed factors (treatment group, sex, weight, and baseline hemoglobin level (80–94 g/L vs. 95–110 g/L). The method of unrestricted least significant differences (LSD) will be applied to ANCOVA results with LS mean values from 95% CI for mean values calculated by the method of least squares for differences between the studied groups. Due to the obvious dependence of the covariates and the base hemoglobin factor (80–94 g/L compared to 95–110 g/L), a linear model containing the term of interaction between these variables will be used.

Non-inferiority will be confirmed if the upper bound of a two-sided confidence interval for the mean value calculated by the method of least squares does not exceed the predetermined non-inferiority margin of 5 g/L. The CI percentage will be determined by the moment of the analysis (interim/final) in accordance with clause 2.3 of the Statistical Analysis Plan.

#### 8.2. Analysis of the secondary endpoint

/Logotype: Research/

- Absolute values and changes in hemoglobin level (g/L) after 4, 8, and 12 weeks of therapy (determined at the final visit) between the study groups.
- Changes in iron metabolism parameters mean values (ferritin, transferrin, percent transferrin saturation, serum iron) during the therapy period (from the screening to the study end visit) in the study groups.
- The responder rate (%) was determined as an increase in the hemoglobin level by  $\geq 20$  g/L after 12 weeks of treatment (from screening to the study end visit) in the study groups.

The data will be checked for compliance with the normal distribution law using the Shapiro-Wilk test.

Intergroup comparison of secondary endpoints related to quantitative scales will be performed using Student's t-test for independent samples if the data correspond to the normal distribution law; otherwise, the Mann–Whitney U test will be applied to independent samples.

Intergroup comparisons of secondary endpoints related to categorical scales will be performed using Pearson's chi-square test if the number of points in each cell of the crosstab is  $\geq 5$ , or Fisher's exact test if at least one of the crosstab cells contains < 5 points.

The dynamics will be assessed using ANOVA methods with repeated measurements if the data correspond to the normal distribution; otherwise, the Friedman test will be applied.

### STATISTICAL ANALYSIS PLAN

#### 9. Safety analysis

Safety evaluation of the study therapy will be performed throughout the study and will be based on the detection of any adverse events occurring during the study. The following will be performed:

- Physical examination, including measurement of blood pressure and heart rate, and gastrointestinal disorders identification (at the screening, during the second visit, and the final visit).
- Complete blood count (at screening and in 4, 8, and 12 weeks of treatment);
- Blood biochemistry (at screening and after 12 weeks of treatment);
- Clinical urinalysis, pregnancy test (at screening and in 12 weeks);
- Registration of concomitant therapy (at each visit).

#### 9.1. Adverse events

The safety assessment will include determining the total number, frequency, and severity of:

- 1. Adverse events (AEs), regardless of their relation to the treatment;
- 2. AEs associated or potentially associated with the medicinal product;
- 3. AEs requiring treatment discontinuation.

Adverse events will be coded using the MedDRA nomenclature in the latest version. These will be represented by the preferred term (PT) and systemic organ class (SOC).

Methods of descriptive statistics will be used to represent the results. Comparison of the incidence of new cases of AE in the study groups will be carried out using Fisher's exact test or Pearson's  $\chi^2$  test, depending on the number of observations in one cell (< 5 or  $\geq$  5).

Changes in the results of laboratory tests over time and the incidence of abnormal test results (based on the reference values of the central laboratory) will be summarized by groups, and a comparison will be made between the groups using appropriate tests for quantitative and qualitative data.

Safety data will be analyzed using the methods designated for the application of efficacy data evaluation.

### STATISTICAL ANALYSIS PLAN

#### 9.2. Other safety endpoints

No other safety endpoints are foreseen in this study.

#### 10. Exploratory analysis

In the course of this study, exploratory analysis is not envisaged.

#### 11. **Interim analysis**

One interim analysis is planned to assess the primary and secondary efficacy endpoints when a group of patients with available data on the primary endpoint will include at least 200 subjects [100 patients in each treatment group: in the main treatment group of patients taking Ferrum Lek® (iron (III) hydroxide polymaltosate complex) and in the control group of patients taking MALTOFER® (iron (III) hydroxide polymaltosate complex]. Safety and efficacy will be assessed in all patients who have received at least one dose of randomized therapy at the time of the interim analysis. Based on the results of the interim analysis of the primary and secondary statistical endpoints of efficacy and safety, the Sponsor may decide to discontinue the study if the endpoints of the study are achieved in accordance with the protocol based on the results of the interim analyses or the sample size can be recalculated using the results of the interim analysis.

| /Logotyne: | Reasearch/ |
|------------|-------------|
| LUZULYPC. | Treuseuren/ |

## STATISTICAL ANALYSIS PLAN

## **Appendix 1. Table layouts**

#### PRIMARY ENDPOINT

| Parameter | Coef. | Standard error | <i>t</i> -value | <i>p</i> -value | C | I |
|---|---|---|---|---|---|---|
| Constant (intercept) | | | | | | |
| Group R versus Group T | | | | | | |
| Gender M versus F | | | | | | |
| Weight | | | | | | |
| Base hemoglobin factor (80–94 g/L compared to 95–110 g/L) | | | | | | |
| Hemoglobin level at screening | | | | | | |
| Interactions | | | | | | |

## STATISTICAL ANALYSIS PLAN

### SECONDARY ENDPOINTS

Table 1. Hemoglobin, frequency analysis of the treatment efficacy after 12 weeks

| Hemoglobin (g/L) | | |
|---|---|---|
| Group | Parameter | Value |
| | Total observations | |
| R – Maltofer <sup>®</sup> | Responders, n | |
| | Responders, % | |
| | 95% CI | |
| | Total observations | |
| T – Ferrum Lek® | Responders, n | |
| 1 1 3 1 | Responders, % | |
| | 95% CI | |
| Group comparison | Pearson's chi-square test, p-value | |

Table 2. Results of analysis of variance

| Coefficients | Evaluation | Standard error | t-value | p-value |
|---|---|---|---|---|
| (Intercept) | | | | |
| V1_CB_LBORRES_HB | | | | |
| (Hemoglobin level at screening) | | | | |
| Group T – Ferrum Lek® | | | | |
| (Test to reference group factor) | | | | |

Table 3. Hemoglobin, absolute values, g/L

| Hemoglobin (g/L) | | | | | |
|---|---|---|---|---|---|
| Group | Parameter | Screening | Week 4 | Week 8 | Week 12 |
| | Number of observations | | | | |
| | Number of missing values | | | | |
| | Mean value | | | | |
| R – Maltofer® | 95% CI | | | | |
| K – Manorci | Standard deviation | | | | |
| | Median | | | | |
| | Minimum value | | | | |
| | Maximum value | | | | |

| | | | 1 |
|-----------------|--------------------------------|------|------|
| | 1st quartile | | |
| | 3rd quartile | | |
| | Interquartile range | | |
| | p-value<br>(Shapiro–Wilk test) | | |
| | Number of observations | | |
| | Number of missing values | | |
| | Mean value | | |
| | 95% CI | | |
| | Standard deviation | | |
| | Median | | |
| T – Ferrum Lek® | Minimum value | | |
| | Maximum value | | |
| | 1st quartile | | |
| | 3rd quartile | | |
| | Interquartile range | | |
| | p-value<br>(Shapiro–Wilk test) | | |
| Group | Criterion | <br> | <br> |
| comparison | p-value | | |
| comparison | p-value | | |

Table 4. Hemoglobin, changes, g/L

| Hemoglobin (g/L) | | | | |
|---|---|---|---|---|
| Group | Parameter | Week 4 – Screening | Week 8 – Screening | Week 12 – Screening |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| R – Maltofer® | Minimum value | | | |
| | Maximum value | | | |
| | 1st quartile | | | |
| | 3rd quartile | | | |
| | Interquartile range | | | |
| | p-value<br>(Shapiro–Wilk test) | | | |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| T – Ferrum Lek® | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| | Minimum value | | | |

| | Maximum value |
|------------------|--------------------------------|
| | 1st quartile |
| | 3rd quartile |
| | Interquartile range |
| | p-value<br>(Shapiro–Wilk test) |
| Group comparison | Criterion |
| | p-value |

Table 5. Blood serum iron, absolute values,  $\mu$ mol/L

| | Serum iron level (µmol/L) | | | | |
|---|---|---|---|---|---|
| Group | Parameter | Screening | Week 4 | Week 8 | Week 12 |
| | Number of observations | | | | |
| | Number of missing values | | | | |
| | Mean value | | | | |
| R – Maltofer® | 95% CI | | | | |
| K – Manorei | Standard deviation | | | | |
| | Median | | | | |
| | Minimum value | | | | |
| | Maximum value | | | | |

| | | T | | , |
|---|---|---|---|---|
| 1st quartile | | | | |
| 3rd quartile | | | | |
| Interquartile range | | | | |
| p-value<br>(Shapiro–Wilk test) | | | | |
| Number of observations | | | | |
| Number of missing values | | | | |
| Mean value | | | | |
| 95% CI | | | | |
| Standard deviation | | | | |
| Median | | | | |
| Minimum value | | | | |
| Maximum value | | | | |
| 1st quartile | | | | |
| 3rd quartile | | | | |
| Interquartile range | | | | |
| p-value<br>(Shapiro–Wilk test) | | | | |
| Criterion | | | | |
| p-value | | | | |
| | Interquartile range p-value (Shapiro-Wilk test) Number of observations Number of missing values Mean value 95% CI Standard deviation Median Minimum value Ist quartile 3rd quartile Interquartile range (Shapiro-Wilk test) Criterion | Interquartile range p-value (Shapiro-Wilk test) Number of observations Number of missing values Mean value 95% CI Standard deviation Median Minimum value Ist quartile 3rd quartile Interquartile range p-value (Shapiro-Wilk test) Criterion | 3rd quartile Interquartile range p-value (Shapiro-Wilk test) Number of observations Number of missing values Mean value 95% CI Standard deviation Median Minimum value Ist quartile 3rd quartile Interquartile range (Shapiro-Wilk test) Criterion | 3rd quartile Interquartile range p-value (Shapiro-Wilk test) Number of observations Number of missing values Mean value 95% CI Standard deviation Median Minimum value 1st quartile 3rd quartile Interquartile range p-value (Shapiro-Wilk test) Criterion |

Table 6. Blood serum iron, changes,  $\mu$ mol/L

| Serum iron level (µmol/L) | | | | |
|---|---|---|---|---|
| Group | Parameter | Week 4 –<br>Screening | Week 8 –<br>Screening | Week 12 –<br>Screening |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| $R-Maltofer^{\mathbb{R}}$ | Minimum value | | | |
| | Maximum value | | | |
| | 1st quartile | | | |
| | 3rd quartile | | | |
| | Interquartile range | | | |
| | p-value<br>(Shapiro–Wilk test) | | | |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| $T-Ferrum\ Lek^{\circledast}$ | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| | Minimum value | | | |

| | Maximum value |
|------------------|--------------------------------|
| | 1st quartile |
| | 3rd quartile |
| | Interquartile range |
| | p-value<br>(Shapiro–Wilk test) |
| Group comparison | Criterion |
| Group comparison | p-value |

Table 7. Transferrin, absolute values, g/L

| | Transferrin (g/L) | | | | |
|---|---|---|---|---|---|
| Group | Parameter | Screening | Week 4 | Week 8 | Week 12 |
| | Number of observations | | | | |
| | Number of missing values | | | | |
| | Mean value | | | | |
| | 95% CI | | | | |
| | Standard deviation | | | | |
| | Median | | | | |
| R – Maltofer® | Minimum value | | | | |
| | Maximum value | | | | |
| | 1st quartile | | | | |
| | 3rd quartile | | | | |
| | Interquartile range | | | | |
| | p-value (Shapiro–Wilk test) | | | | |
| | Number of observations | | | | |
| | Number of missing values | | | | |
| | Mean value | | | | |
| T – Ferrum Lek® | 95% CI | | | | |
| | Standard deviation | | | | |
| | Median | | | | |

| | Minimum value |
|---------------------|-----------------------------|
| | Maximum value |
| | 1st quartile |
| | 3rd quartile |
| | Interquartile range |
| | p-value (Shapiro–Wilk test) |
| Group<br>comparison | Criterion |
| | p-value |

Table 8. Transferrin, changes, g/L

| | Transferrin (g/L) | | | |
|---|---|---|---|---|
| Group | Parameter | Week 4 – Screening | Week 8 – Screening | Week 12 – Screening |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| R – Maltofer® | Minimum value | | | |
| | Maximum value | | | |
| | 1st quartile | | | |
| | 3rd quartile | | | |
| | Interquartile range | | | |
| | p-value<br>(Shapiro–Wilk test) | | | |
| | Number of observations | | | |
| | Number of missing values | | | |
| T – Ferrum Lek® | Mean value | | | |
| 1 - 1 Cituili LCK | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |

| | Minimum value |
|------------------|--------------------------------|
| | Maximum value |
| | 1st quartile |
| | 3rd quartile |
| | Interquartile range |
| | p-value<br>(Shapiro–Wilk test) |
| Group comparison | Criterion |
| | p-value |

Table 9. Percentage of transferrin saturation with iron, absolute values (%)

| Percentage of transferrin saturation with iron (%) | | | | | |
|---|---|---|---|---|---|
| Group | Parameter | Screening | Week 4 | Week 8 | Week 12 |
| | Number of observations | | | | |
| | Number of missing values | | | | |
| | Mean value | | | | |
| D. M.I. C. R | 95% CI | | | | |
| R – Maltofer® | Standard deviation | | | | |
| | Median | | | | |
| | Minimum value | | | | |
| | Maximum value | | | | |

| T | 1 | 1 | 1 | 1 |
|------------------|--------------------------------|---|---|---|
| | 1st quartile | | | |
| | 3rd quartile | | | |
| | Interquartile range | | | |
| | p-value<br>(Shapiro–Wilk test) | | | |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| T – Ferrum Lek® | Minimum value | | | |
| | Maximum value | | | |
| | 1st quartile | | | |
| | 3rd quartile | | | |
| | Interquartile range | | | |
| | p-value<br>(Shapiro–Wilk test) | | | |
| Crown or | Criterion | | | |
| Group comparison | p-value | | | |

Table 10. Percentage of transferrin saturation with iron, changes (%)

| Percentage of transferrin saturation with iron (%) | | | |
|---|---|---|---|
| Group | Parameter | Week 4 – Week 8 Screening Screening | Week 12 –<br>Screening |
| | Number of observations | | |
| | Number of missing values | | |
| | Mean value | | |
| | 95% CI | | |
| | Standard deviation | | |
| | Median | | |
| $R-Maltofer^{\circledR}$ | Minimum value | | |
| | Maximum value | | |
| | 1st quartile | | |
| | 3rd quartile | | |
| | Interquartile range | | |
| | p-value (Shapiro–Wilk test) | | |
| | Number of observations | | |
| | Number of missing values | | |
| T – Ferrum Lek® | Mean value | | |
| 1 – I cituiii Lek | 95% CI | | |
| | Standard deviation | | |
| | Median | | |

| | Minimum value |
|------------------|-----------------------------|
| | Maximum value |
| | 1st quartile |
| | 3rd quartile |
| | Interquartile range |
| | p-value (Shapiro–Wilk test) |
| Group comparison | Criterion |
| Group comparison | p-value |
Table 11. Ferritin, absolute values,  $\mu g/L$ 

| | Serun | n ferritin level (μ | g/L) | | |
|---|---|---|---|---|---|
| Group | Parameter | Screening | Week 4 | Week 8 | Week 12 |
| | Number of observations | | | | |
| | Number of missing values | | | | |
| | Mean value | | | | |
| | 95% CI | | | | |
| | Standard deviation | | | | |
| | Median | | | | |
| R – Maltofer® | Minimum value | | | | |
| | Maximum value | | | | |
| | 1st quartile | | | | |
| | 3rd quartile | | | | |
| | Interquartile range | | | | |
| | p-value<br>(Shapiro–Wilk test) | | | | |
| | Number of observations | | | | |
| T – Ferrum Lek® | Number of missing values | | | | |
| | Mean value | | | | |
| | 95% CI | | | | |

| | | | T |
|------------------|--------------------------------|------|------|
| | Standard deviation | | |
| | Median | | |
| | Minimum value | | |
| | Maximum value | | |
| | 1st quartile | | |
| | 3rd quartile | | |
| | Interquartile range | | |
| | p-value<br>(Shapiro–Wilk test) | | |
| Group comparison | Criterion | <br> | <br> |
| oup companion | p-value | | |

Table 12. Ferritin, changes,  $\mu g/L$ 

| | Serum ferritin level (μg/L) | | | |
|---|---|---|---|---|
| Group | Parameter | Week 4 –<br>Screening | Week 8 –<br>Screening | Week 12 –<br>Screening |
| | Number of observations | | | |
| | Number of missing values | | | |
| | Mean value | | | |
| | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |
| $R-Maltofer^{\circledR}$ | Minimum value | | | |
| | Maximum value | | | |
| | 1st quartile | | | |
| | 3rd quartile | | | |
| | Interquartile range | | | |
| | p-value<br>(Shapiro–Wilk test) | | | |
| | Number of observations | | | |
| | Number of missing values | | | |
| T – Ferrum Lek® | Mean value | | | |
| 1 – 1 ciruiii Lek | 95% CI | | | |
| | Standard deviation | | | |
| | Median | | | |

| | Minimum value |
|------------------|-----------------------------|
| | Maximum value |
| | 1st quartile |
| | 3rd quartile |
| | Interquartile range |
| | p-value (Shapiro–Wilk test) |
| Group comparison | Criterion |
| Group comparison | p-value |

### STATISTICAL ANALYSIS PLAN

#### LABORATORY RESULTS

Table 1. Urinalysis

| Visit | Group | Parameter | рН | Protein | Specific gravity | RBC |
|---|---|---|---|---|---|---|
| | | N | | | | |
| | | Missed | | | | |
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |
| | | 95% CI | | | | |
| | Treatment group: $R - Maltofer^{$ ® | SD | | | | |
| | K – Manoter | Median | | | | |
| V1 | | Min | | | | |
| V I | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |
| | | N | | | | |
| | Treatment group:<br>T – Ferrum Lek® | Missed | | | | |
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |

| Visit | Group | Parameter | рН | Protein | Specific gravity | RBC |
|---|---|---|---|---|---|---|
| | | 95% CI | | | | |
| | | SD | | | | |
| | | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |
| | | N | | | | |
| | | Missed | | | | |
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |
| | | 95% CI | | | | |
| | Treatment group: $R - Maltofer^{$ ® | SD | | | | |
| V5 | K – Waltolei | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |
| | | N | | | | |

| Visit | Group | Parameter | pН | Protein | Specific gravity | RBC |
|---|---|---|---|---|---|---|
| | | Missed | | | | |
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |
| | | 95% CI | | | | |
| | Treatment group: | SD | | | | |
| | T – Ferrum Lek® | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |

Table 2. Urinalysis statistical test

| Vis | sit | V1 | V5 | V1 | V5 | V1 | V5 | V1 | V5 |
|---|---|---|---|---|---|---|---|---|---|
| Varia | able | p | Н | Pro | tein | Specific | gravity | RI | 3C |
| Shapira Wills tast n value | Treatment group: $R - Maltofer^{$ ® | | | | | | | | |
| Shapiro–Wilk test, p-value | Treatment group: T – Ferrum Lek® | | | | | | | | |
| Student's t-te | est, p-value | | | | | | | | |
| Wilcoxon-Mann-W | hitney test, p-value | | | | | | | | |

### STATISTICAL ANALYSIS PLAN

Table 3. Urinalysis, categorical variables

| Visit | Variable | Group | Distribution of responses | Chi-square test, p-value |
|---|---|---|---|---|
| | WDG | Treatment group:<br>R – Maltofer® | | |
| 3/1 | WBC | Treatment group:<br>T – Ferrum Lek® | | |
| V1 | C.L. | Treatment group: R – Maltofer® | | |
| | Color | Treatment group:<br>T – Ferrum Lek® | | |
| | WDC | Treatment group:<br>R – Maltofer® | | |
| 7/5 | WBC | Treatment group: T – Ferrum Lek® | | |
| V5 | 6.1 | Treatment group: R – Maltofer® | | |
| | Color | Treatment group:<br>T – Ferrum Lek® | | |

Table 4. Hematology 1

| Visit | Group | Parameter | Hematocrit (%) | Hemoglobin | RBC |
|---|---|---|---|---|---|
| | | N | | | |
| | Treatment groups | Missed | | | |
| V1 | Treatment group: R – Maltofer® | Beyond the limit of detection | | | |
| | | Mean | | | |

| Visit | Group | Parameter | Hematocrit (%) | Hemoglobin | RBC |
|---|---|---|---|---|---|
| | | 95% CI | | | |
| | | SD | | | |
| | | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | Treatment group: | SD | | | |
| | T – Ferrum Lek® | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| V3 | Treatment group: | N | | | |
| V 3 | R – Maltofer® | Missed | | | |

| Visit | Group | Parameter | Hematocrit (%) | Hemoglobin | RBC |
|---|---|---|---|---|---|
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | | SD | | | |
| | | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | Treatment group: | 95% CI | | | |
| | Treatment group:<br>T – Ferrum Lek® | SD | | | |
| | | Median | | | |
| | | Min | | | |
| | | Max | · | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |

| Visit | Group | Parameter | Hematocrit (%) | Hemoglobin | RBC |
|---|---|---|---|---|---|
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | Treatment group: $R - Maltofer^{$ ® | SD | | | |
| | K – Manorer | Median | | | |
| | | Min | | | |
| | | Max | | | |
| V4 | | Q1.25% | | | |
| V 4 | | Q3.75% | | | |
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | Treatment group:<br>T – Ferrum Lek® | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | | SD | | | |
| | | Median | | | |
| | | Min | | | |

| Visit | Group | Parameter | Hematocrit (%) | Hemoglobin | RBC |
|---|---|---|---|---|---|
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | Treatment group: $R - Maltofer^{\otimes}$ | SD | | | |
| | K – Manorei | Median | | | |
| | | Min | | | |
| V5 | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| | Treatment group:<br>T – Ferrum Lek® | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |

### STATISTICAL ANALYSIS PLAN

| Visit | Group | Parameter | Hematocrit (%) | Hemoglobin | RBC |
|-------|-------|-----------|----------------|------------|-----|
| | | SD | | | |
| | | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |

Table 5. Hematology 2

| Visit | Group | Parameter | WBC | Lymphocytes | Lymphocytes (%) |
|---|---|---|---|---|---|
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| V1 | Treatment group: R – Maltofer® | SD | | | |
| | K – Manorei | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |

### STATISTICAL ANALYSIS PLAN

| Visit | Group | Parameter | WBC | Lymphocytes | Lymphocytes (%) |
|---|---|---|---|---|---|
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | Treatment group:<br>T – Ferrum Lek® | SD | | | |
| | 1 – Feffulli Lek | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |

Table 6. Hematology 3

| Visit | Group | Parameter | Neutrophils | Neutrophils (%) | Stab neutrophils (%) | Segmented neutrophils (%) |
|---|---|---|---|---|---|---|
| | | N | | | | |
| | | Missed | | | | |
| | Treatment aroun. | Beyond the limit of | | | | |
| V1 | Treatment group: R – Maltofer® | detection | | | | |
| | K – Maitolei | Mean | | | | |
| | | 95% CI | | | | |
| | | SD | | | | |

| Visit | Group | Parameter | Neutrophils | Neutrophils (%) | Stab neutrophils (%) | Segmented neutrophils (%) |
|---|---|---|---|---|---|---|
| | | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |
| | | N | | | | |
| | | Missed | | | | |
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |
| | | 95% CI | | | | |
| | Treatment group:<br>T – Ferrum Lek® | SD | | | | |
| | 1 – Ferrum Lek | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |

### STATISTICAL ANALYSIS PLAN

Table 7. Hematology 4

| Visit | Group | Parameter | Basophils | Basophils (%) | ESR | Platelets | Eosinophils | Eosinophils (%) |
|---|---|---|---|---|---|---|---|---|
| | | N | | | | | | |
| | | Missed | | | | | | |
| | | Beyond the limit of detection | | | | | | |
| | | Mean | | | | | | |
| | Tuester out answer | 95% CI | | | | | | |
| | Treatment group: $R - Maltofer^{\mathbb{R}}$ | SD | | | | | | |
| | | Median | | | | | | |
| | | Min | | | | | | |
| V1 | | Max | | | | | | |
| <b>V</b> 1 | | Q1.25% | | | | | | |
| | | Q3.75% | | | | | | |
| | | IQR.75% | | | | | | |
| | | N | | | | | | |
| | | Missed | | | | | | |
| | Treatment group: T – Ferrum Lek® | Beyond the limit of detection | | | | | | |
| | | Mean | | | | | | |
| | | 95% CI | | | | | | |
| | | SD | | | | | | |

| Visit | Group | Parameter | Basophils | Basophils (%) | ESR | Platelets | Eosinophils | Eosinophils (%) |
|---|---|---|---|---|---|---|---|---|
| | | Median | | | | | | |
| | | Min | | | | | | |
| | | Max | | | | | | |
| | | Q1.25% | | | | | | |
| | | Q3.75% | | | | | | |
| | | IQR.75% | | | | | | |

### STATISTICAL ANALYSIS PLAN

Table 8. Hematology, statistical test 1

| remaiology, sta | tibiledii test 1 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Vi | isit | V1 | V3 | V4 | V5 | V1 | V3 | V4 | V5 | V1 | V3 | V4 | V5 |
| Vari | iable | | Hemato | ocrit (%) | | | Hemo | globin | | | RI | BC | |
| Shapiro- | Treatment<br>group: R –<br>Maltofer® | | | | | | | | | | | | |
| Wilk test, p-<br>value | Treatment<br>group: T –<br>Ferrum Lek® | | | | | | | | | | | | |
| Student's t-t | test, p-value | | | | | | | | | | | | |
| | –Whitney test, p-lue | | | | | | | | | | | | |

Table 9. Hematology, statistical test 2

| Vi | sit | V1 | | |
|---|---|---|---|---|
| Vari | able | WBC | Lymphocytes | Lymphocytes (%) |
| Shapiro– | Treatment group: R – Maltofer® | | | |
| Wilk test, p-value | Treatment group:<br>T – Ferrum Lek® | | | |
| Student's t- | | | | |
| Wilcoxon-Mann-W | Whitney test, p-value | | | |

Table 10. Hematology, statistical test 3

| Visit | V1 |
|-------|----|
|-------|----|

### STATISTICAL ANALYSIS PLAN

| Variable | | Neutrophils | Neutrophils (%) | Stab neutrophils (%) | Segmented neutrophils (%) |
|---|---|---|---|---|---|
| Shapiro- | Treatment group: R – Maltofer® | | | | |
| Wilk test, p-value | Treatment group:<br>T – Ferrum Lek® | | | | |
| Student's t-test, p-value | | | | | |
| Wilcoxon-Mann-W | hitney test, p-value | | | | |

Table 11. Hematology, statistical test 4

| V | Visit | | | V1 | | | |
|---|---|---|---|---|---|---|---|
| Variable | | Basophils | Basophils (%) | ESR | Platelets | Eosinophils | Eosinophils (%) |
| Chanina Wills test a value | Treatment group: R – Maltofer® | | | | | | |
| Shapiro–Wilk test, p-value | Treatment group:<br>T – Ferrum Lek <sup>®</sup> | | | | | | |
| Student's t-test, p-value | | | | | | | |
| Wilcoxon-Mann-V | Whitney test, p-value | | | | | | |

Table 12. Physiological data

| Visit | Group | Parameter | Weight | Age | BMI | Height |
|------------------|---------------|-----------|--------|-----|-----|--------|
| Treatment group: | N | | | | | |
| V I | R – Maltofer® | Missed | | | | |

| Visit | Group | Parameter | Weight | Age | BMI | Height |
|---|---|---|---|---|---|---|
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |
| | | 95% CI | | | | |
| | | SD | | | | |
| | | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |
| | | IQR.75% | | | | |
| | | N | | | | |
| | | Missed | | | | |
| | | Beyond the limit of detection | | | | |
| | | Mean | | | | |
| | Treatment group: | 95% CI | | | | |
| | T – Ferrum Lek® | SD | | | | |
| | | Median | | | | |
| | | Min | | | | |
| | | Max | | | | |
| | | Q1.25% | | | | |
| | | Q3.75% | | | | |

### STATISTICAL ANALYSIS PLAN

| Visit | Group | Parameter | Weight | Age | BMI | Height |
|-------|-------|-----------|--------|-----|-----|--------|
| | | IQR.75% | | | | |

Table 13. Physiological data, statistical test

| The state of the s | Visit | | | V1 | |
|---|---|---|---|---|---|
| Va | riable | Weight | Age | BMI | Height |
| Shapiro– | Treatment group: R – Maltofer® | | | | |
| Wilk test, p-value | Treatment group:<br>T – Ferrum Lek <sup>®</sup> | | | | |
| Student's t | Student's t-test, p-value | | | | |
| Wilcoxon-Mann- | Wilcoxon-Mann-Whitney test, p-value | | | | |

Table 14. Physiological data, categorical data

| Visit | Variable | Group | Distribution of responses | Chi-square test, p-value |
|---|---|---|---|---|
| V1 | Condon | Treatment group: R – Maltofer® | | |
| V1 | Gender | Treatment group:<br>T – Ferrum Lek® | | |

Table 15. Biochemistry 1

| Visit | Group | Parameter | ALT | AST | Total protein | Total bilirubin | C-reactive protein |
|---|---|---|---|---|---|---|---|
| V1 | Treatment group: | N | | | | | |
| | R – Maltofer® | Missed | | | | | |

| Visit | Group | Parameter | ALT | AST | Total protein | Total bilirubin | C-reactive protein |
|---|---|---|---|---|---|---|---|
| | | Beyond the limit of detection | | | | | |
| | | Mean | | | | | |
| | | 95% CI | | | | | |
| | | SD | | | | | |
| | | Median | | | | | |
| | | Min | | | | | |
| | | Max | | | | | |
| | | Q1.25% | | | | | |
| | | Q3.75% | | | | | |
| | | IQR.75% | | | | | |
| | | N | | | | | |
| | | Missed | | | | | |
| | | Beyond the limit of detection | | | | | |
| | | Mean | | | | | |
| | Treatment group:<br>T – Ferrum Lek® | 95% CI | | | | | |
| | I – Ferrum Lek® | SD | | | | | |
| | | Median | | | | | |
| | | Min | | | | | |
| | | Max | | | | | |
| | | Q1.25% | | | | | |

| Visit | Group | Parameter | ALT | AST | Total protein | Total bilirubin | C-reactive protein |
|---|---|---|---|---|---|---|---|
| | | Q3.75% | | | | | |
| | | IQR.75% | | | | | |
| | | N | | | | | |
| | | Missed | | | | | |
| | | Beyond the limit of detection | | | | | |
| | | Mean | | | | | |
| | | 95% CI | | | | | |
| | Treatment group: $R - Maltofer^{\otimes}$ | SD | | | | | |
| | K – Manoier | Median | | | | | |
| | | Min | | | | | |
| 375 | | Max | | | | | |
| V5 | | Q1.25% | | | | | |
| | | Q3.75% | | | | | |
| | | IQR.75% | | | | | |
| | | N | | | | | |
| | | Missed | | | | | |
| | Treatment group: | Beyond the limit of detection | | | | | |
| | T – Ferrum Lek® | Mean | | | | | |
| | | 95% CI | | | | | |
| | | SD | | | | | |

# STATISTICAL ANALYSIS PLAN

| Visit | Group | Parameter | ALT | AST | Total protein | Total bilirubin | C-reactive protein |
|---|---|---|---|---|---|---|---|
| | | Median | | | | | |
| | | Min | | | | | |
| | | Max | | | | | |
| | | Q1.25% | | | | | |
| | | Q3.75% | | | | | |
| | | IQR.75% | | | | | |

Table 16. Biochemistry 2

| Visit | Group | Parameter | Conjugated bilirubin | Creatinine level | Alkaline phosphatase |
|---|---|---|---|---|---|
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | Treatment group: | 95% CI | | | |
| 7.71 | | SD | | | |
| V1 | $R-Maltofer^{\mathbb{R}}$ | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |

| Visit | Group | Parameter | Conjugated bilirubin | Creatinine level | Alkaline phosphatase |
|---|---|---|---|---|---|
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | Treatment group: T – Ferrum Lek® | SD | | | |
| | I – Ferrum Lek® | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| V5 | Treatment group: $R - Maltofer^{\mathbb{R}}$ | Mean | | | |
| | K – Maitoier | 95% CI | | | |
| | | SD | | | |
| | | Median | | | |
| | | Min | | | |

### STATISTICAL ANALYSIS PLAN

| Visit | Group | Parameter | Conjugated bilirubin | Creatinine level | Alkaline phosphatase |
|---|---|---|---|---|---|
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |
| | | N | | | |
| | | Missed | | | |
| | | Beyond the limit of detection | | | |
| | | Mean | | | |
| | | 95% CI | | | |
| | Treatment group: | SD | | | |
| | T – Ferrum Lek® | Median | | | |
| | | Min | | | |
| | | Max | | | |
| | | Q1.25% | | | |
| | | Q3.75% | | | |
| | | IQR.75% | | | |

Table 17. Biochemistry 3

| Visit | Group | Parameter | T4 | Vitamin B12 | Creatinine index | TSH | Folic acid (B9) |
|---|---|---|---|---|---|---|---|
| V1 | Treatment group: | N | | | | | |
| V I | $R-Maltofer^{\mathbb{R}}$ | Missed | | | | | |

| Visit | Group | Parameter | Т4 | Vitamin B12 | Creatinine index | TSH | Folic acid (B9) |
|---|---|---|---|---|---|---|---|
| | | Beyond the limit of detection | | | | | |
| | | Mean | | | | | |
| | | 95% CI | | | | | |
| | | SD | | | | | |
| | | Median | | | | | |
| | | Min | | | | | |
| | | Max | | | | | |
| | | Q1.25% | | | | | |
| | | Q3.75% | | | | | |
| | | IQR.75% | | | | | |
| | | N | | | | | |
| | | Missed | | | | | |
| | | Beyond the limit of detection | | | | | |
| | | Mean | | | | | |
| | Treatment group:<br>T – Ferrum Lek® | 95% CI | | | | | |
| | I − Ferrum Lek® | SD | | | | | |
| | | Median | | | | | |
| | | Min | | | | | |
| | | Max | | | | | |
| | | Q1.25% | | | | | |

### STATISTICAL ANALYSIS PLAN

| Visit | Group | Parameter | T4 | Vitamin B12 | Creatinine index | TSH | Folic acid (B9) |
|---|---|---|---|---|---|---|---|
| | | Q3.75% | | | | | |
| | | IQR.75% | | | | | |

Table 18. Biochemistry, statistical test 1

| Vi | sit | V1 | V5 | V1 | V5 | V1 | V5 | V1 | V5 | V1 | V5 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Vari | able | AI | LT | A | ST | Total 1 | protein | Total b | ilirubin | ubin C-reactive protein | |
| Shapiro- | Treatment group: R – Maltofer® | | | | | | | | | | |
| Wilk test, p-value | Treatment group:<br>T – Ferrum Lek® | | | | | | | | | | |
| Student's t-test, p-value | | | | | | | | | | | |
| Wilcoxon-Mann-W | hitney test, p-value | | | | | | | | | | |

Table 19. Biochemistry, statistical test 2

| Visit | | V1 | V5 | V1 | V5 | V1 | V5 |
|---|---|---|---|---|---|---|---|
| Variable | | Conjugated bilirubin | | Creatinine level | | Alkaline phosphatase | |
| Shapiro- | Treatment group:<br>R – Maltofer® | | | | | | |
| Wilk test, p-value | Treatment group:<br>T – Ferrum Lek® | | | | | | |
| Student's t-test, p-value | | | | | | | |
| Wilcoxon-Mann-V | Vhitney test, p-value | | | | | | |

| /Logotype: | Reasearch/ |
|------------|--------------|
| LUZULYPU. | Itcuscui cii |

# STATISTICAL ANALYSIS PLAN

Table 20. Biochemistry, statistical test 3

| Vi | Visit | | | V1 | | |
|---|---|---|---|---|---|---|
| , | V ISIV | | | T | | |
| Var | iable | T4 | Vitamin B12 | Creatinine index | TSH | Folic acid (B9) |
| Shapiro- | Treatment group:<br>R – Maltofer <sup>®</sup> | | | | | |
| Wilk test, p-value | Treatment group:<br>T – Ferrum Lek® | | | | | |
| Student's t-test, p-value | | | | | | |
| Wilcoxon-Mann-V | Wilcoxon-Mann-Whitney test, p-value | | | | | |

### STATISTICAL ANALYSIS PLAN

#### **ADVERSE EVENTS**

Table 1. Adverse events reported in the study

| Adverse events | Group | Amount | % of the total number of AEs | % of the number of AEs by the medicinal product | p-value, Fisher's test |
|---|---|---|---|---|---|
| All adverse events | T | | | | |
| An adverse events | R | | | | |
| SOC | T | | | | |
| 500 | R | | | | |
| PT | Т | | | | |
| 11 | R | | | | |
| PT | Т | | | | |
| 11 | R | | | | |
| | Т | | | | |
| | R | | | | |
| SOC | Т | | | | |
| 500 | R | | | | |
| PT | Т | | | | |
| 11 | R | | | | |
| PT | Т | | | | |
| 11 | R | | | | |
| | Т | | | | |
| | R | | | | |

#### STATISTICAL ANALYSIS PLAN

Tables N. Is the adverse event ongoing?/ Relatedness to the medicinal product/ Dose adjustment or temporary withdrawal of the IMP/ Complete withdrawal of the IMP/ Prescribing a concomitant medicinal product/ Prescribing non-drug therapy/ Patient admission to hospital or hospitalization prolongation/ Based on an AE/ Is it an SAE?/ Leads to death/ Threatens life/ Requires admission to hospital or hospitalization prolongation/ Leads to permanent or significant incapacity for work or disability

| Adverse events | Group | {variable name] | Amount | % of the number of AEs by the medicinal product | p-value, Fisher's test |
|---|---|---|---|---|---|
| | | value | | | |
| | T | value | | | |
| A 11 - 1 | | value | | | 1 |
| All adverse events | | value | | | 1 |
| | R | value | | | |
| | | value | | | |
| | | value | | | |
| | T | value | | | 1 |
| SOC | | value | | | |
| SOC | | value | | | |
| | R | value | | | |
| | | value | | | |
| | | value | | | |
| | T | value | | | |
| DT | | value | | | |
| P1 | PT | value | | | 1 |
| | R | value | | | |
| | | value | | | |

| Adverse events | Group | {variable name] | Amount | % of the number of AEs by the medicinal product | p-value, Fisher's test |
|---|---|---|---|---|---|
| | | value | | | |
| | T | value | | | |
| РТ | | value | | | 1 |
| Г1 | | value | | | 1 |
| | R | value | | | |
| | | value | | | |
| | | value | | | |
| | T | value | | | |
| | | value | | | 1 |
| | | value | | | |
| | R | value | | | |
| | | value | | | |
| | | value | | | |
| | Т | value | | | |
| SOC | | value | | | 1 |
| 50C | | value | | | 1 |
| | R | value | | | |
| | | value | | | |
| | | value | | | |
| DT | Т | value | | | 1 |
| РТ | | value | | | 1 |
| | R | value | | | |

| Adverse events | Group | {variable name] | Amount | % of the number of AEs by the medicinal product | p-value, Fisher's test |
|---|---|---|---|---|---|
| | | value | | | |
| | | value | | | |
| PT | Т | value | | | 1 |
| | | value | | | |
| | | value | | | |
| | R | value | | | |
| | | value | | | |
| | | value | | | |
| | Т | value | | | 1 |
| | | value | | | |
| | | value | | | |
| | R | value | | | |
| | | value | | | |
| | | value | | | |